CLINICAL TRIAL: NCT01970449
Title: A Phase 1 Randomized, Double-blind, Placebo Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of an HIV-1 Vaccine Regimen of DNA Prime and NYVAC Boost With 3 Different HIV-1 Envelope Inserts (Nat-B Env, CON-S Env, and Mosaic Env) in Healthy, HIV-1-uninfected Adults
Brief Title: Evaluating the Safety and Immune Response to Three Different Prime-Boost HIV Vaccine Regimens in Healthy, HIV-Uninfected Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); IPPOX Foundation (Other); Center for HIV/AIDS Vaccine Immunology (CHAVI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 099; 11782 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: study vaccines with Nat-B env insert (Experimental): Participants in this arm will receive DNA Nat-B env vaccine injections on Day 0 and Day 28 followed by NYVAC Nat-B env vaccine injections on Day 84 and Day 164.
  Interventions: Biological: DNA Nat-B env vaccine; Biological: NYVAC Nat-B env vaccine; Device: Biojector 2000® Needle-Free Injection Management System™ (Biojector 2000®)
- Group 1: placebo vaccines with Nat-B env insert (Placebo Comparator): Participants in this arm will receive placebo injections of DNA Nat-B env vaccine on Day 0 and Day 28 followed by placebo injections for NYVAC Nat-B env vaccine on Day 84 and Day 164.
  Interventions: Biological: Placebo
- Group 2: study vaccines with CON-S env insert (Experimental): Participants in this arm will receive DNA CON-S env vaccine injections on Day 0 and Day 28 followed by NYVAC CON-S env vaccine injections on Day 84 and Day 164.
  Interventions: Biological: DNA CON-S env vaccine; Biological: NYVAC CON-S env vaccine; Device: Biojector 2000® Needle-Free Injection Management System™ (Biojector 2000®)
- Group 2: placebo vaccines with CON-S env insert (Placebo Comparator): Participants in this arm will receive placebo injections of DNA CON-S env vaccine on Day 0 and Day 28 followed by placebo injections for NYVAC CON-S env vaccine on Day 84 and Day 164.
  Interventions: Biological: Placebo
- Group 3: study vaccines with Mosaic env insert (Experimental): Participants in this arm will receive DNA Mosaic env vaccine injections on Day 0 and Day 28 followed by NYVAC Mosaic env vaccine injections on Day 84 and Day 164.
  Interventions: Biological: DNA Mosaic env vaccine; Biological: NYVAC Mosaic env vaccine; Device: Biojector 2000® Needle-Free Injection Management System™ (Biojector 2000®)
- Group 3: placebo vaccines with Mosaic env insert (Placebo Comparator): Participants in this arm will receive placebo injections of DNA Mosaic env vaccine on Day 0 and Day 28 followed by placebo injections for NYVAC Mosaic env vaccine on Day 84 and Day 164.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DNA Nat-B env vaccine — The DNA Nat-B env vaccine will be administered as a 4-mg dose injection intramuscularly (IM) by Biojector 2000 ® in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 1: study vaccines with Nat-B env insert
Biological: NYVAC Nat-B env vaccine — NVYAC Nat-B env vaccine will be administered as a 3 × 10^7 plaque forming units (pfu) dose IM by needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 1: study vaccines with Nat-B env insert
Biological: DNA CON-S env vaccine — The DNA CON-S env vaccine will be administered as a 4-mg dose injection IM by Biojector 2000 ® in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 2: study vaccines with CON-S env insert
Biological: NYVAC CON-S env vaccine — NVYAC CON-S env vaccine will be administered as a 3 × 10^7 pfu dose IM by needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 2: study vaccines with CON-S env insert
Biological: DNA Mosaic env vaccine — The DNA Mosaic env vaccine will be administered as a 4-mg dose injection IM by Biojector 2000 ® in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 3: study vaccines with Mosaic env insert
Biological: NYVAC Mosaic env vaccine — NVYAC Mosaic env vaccine will be administered as a 3 × 10^7 pfu dose IM by needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated).
  Arms: Group 3: study vaccines with Mosaic env insert
Biological: Placebo — Placebo for both DNA and NYVAC vaccines will be administered in the deltoid muscle of the non-dominant arm (unless medically contraindicated) as sodium chloride for injection, 0.9%.
  Arms: Group 1: placebo vaccines with Nat-B env insert; Group 2: placebo vaccines with CON-S env insert; Group 3: placebo vaccines with Mosaic env insert
Device: Biojector 2000® Needle-Free Injection Management System™ (Biojector 2000®) — All three DNA env vaccines will be administered IM in the deltoid muscle of the non-dominant arm (unless medically contraindicated) using the Biojector 2000® device.
  Arms: Group 1: study vaccines with Nat-B env insert; Group 2: study vaccines with CON-S env insert; Group 3: study vaccines with Mosaic env insert

SUMMARY:
The purpose of this study is to test the safety and immune response to three different sets of HIV vaccines in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and immune response to three different HIV-1 prime-boost vaccine regimens in healthy, HIV-1-uninfected adults. The regimens will differ by the type of HIV-1 envelope insert (Nat-B env, CON-S env, or Mosaic env) contained in both the DNA prime vaccine and the NYVAC boost vaccine.

The study will enroll 180 healthy, HIV-1-uninfected adults in two stages (Part A and Part B). After Part A of the study is fully enrolled, study researchers will evaluate study immunogenicity data to determine whether to enroll participants into Part B. The study design and vaccination schedule for both parts of the study will be the same.

Participants will be randomly assigned to one of three groups and receive either one of the experimental vaccine regimens or a placebo vaccine regimen. Participants will receive four total injections: on Day 0 and Day 28 (DNA vaccine or placebo) and on Day 84 and Day 168 (NYVAC vaccine or placebo). Group 1 participants will receive DNA Nat-B env and NYVAC Nat-B env vaccines, Group 2 participants will receive DNA CON-S env and NYVAC CON-S env vaccines, and Group 3 participants will receive DNA Mosaic env and NYVAC Mosaic env vaccines.

Total study duration will be either 3 years after enrollment (for participants in the United States) or 5 years after enrollment (for participants in Switzerland). For all participants, study visits will occur on Days 0, 14, 28, 42, 84, 98, 168, 175, 182, 273, 357, and 364. After the last study visit, participants will be contacted annually by phone or e-mail for a total of 3 (U.S. participants) or 5 (Switzerland participants) years to answer questions about their health.

At screening, participants will give a medical history; undergo a complete physical exam, blood collection, urine collection, and an electrocardiogram (ECG); and receive risk reduction counseling. At most follow-up visits, participants will undergo an abbreviated physical exam, blood collection, urine collection, and receive risk reduction counseling. Participants will have additional ECGs on Days 98 and 182. At all visits, female participants who were born female will be assessed for pregnancy prevention, and at select visits, will undergo a pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years for U.S. participants (5 years for participants in Switzerland) following initial study injection
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin greater than or equal to 12.5 g/dL for participants who were born female, or greater than or equal to 13.5 g/dL for participants who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: ALT, AST, and alkaline phosphatase less than 1.25 times the institutional upper limit of normal (ULN); creatinine less than or equal to ULN
* Cardiac Troponin T or I (cTnT or cTnI) does not exceed the institutional ULN
* Negative HIV-1 and -2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay. Non-U.S. sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine: Negative urine glucose, negative or trace urine protein, and negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A participant who was born female must agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; less than or equal to 18; or greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Intent to participate in another study of an investigational research agent during the planned duration of this study
* Pregnant or breastfeeding
* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 099 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis and the identity of the study control/placebo must be obtained.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 099 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 099 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency
* Hypersensitivity to eggs and/or egg products
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension: If a participant has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled (as defined in the protocol). If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment. More information on this criterion can be found in the protocol.
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, or clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* Participants who have 2 or more of the following cardiac risk factors: participant report of history of elevated blood cholesterol defined as fasting LDL greater than 160 mg/dL; first degree relative (e.g., mother, father, brother, or sister) who had coronary artery disease before the age of 50 years; current smoker; or BMI greater than or equal to 35
* ECG with clinically significant findings or features that would interfere with the assessment of myo/pericarditis, as determined by the contract ECG Lab, cardiologist, or study clinician. More information on this criterion can be found in the protocol.
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: Participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of local injection site reactogenicity signs and symptoms | Measured for 3 days following each vaccination visit (Days 0, 28, 84, and 168)
  Local injection site signs and symptoms may include pain, tenderness, erythema, induration, and maximum severity of pain and/or tenderness.
Frequency of adverse events (AEs) categorized by the MedDRA body system, MedDRA preferred term, severity and assessed relationship to study products; detailed description of all AEs meeting DAIDS criteria for expedited reporting (EAE) | Measured through Day 364 visit
  MedDRA is the Medical Dictionary for Regulatory Activities.
Laboratory measures of safety | Measured through Day 357 visit
  Laboratory measures of safety include white blood cells (WBC), neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase (ALT), alkaline phosphatase (ALK Phos), aspartate aminotransferase (AST), and creatinine.
Number of participants with early discontinuation of vaccinations and reason for discontinuation | Measured through Day 364 visit
Breadth of the T-cell response determined as the number of reactive CD4 and CD8 T-cell epitopes using global potential T-cell epitope (PTEg) peptides | Measured through Day 182 visit
Total magnitude of CD4 and CD8 T-cell responses measured by intracellular cytokine staining (ICS) to PTEg peptide pools | Measured through Day 182 visit
Frequency and severity of systemic reactogenicity signs and symptoms | Measured for 3 days following each vaccination visit (Days 0, 28, 84, and 168)
  Systemic reactogenicity signs and symptoms may include fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms.

SECONDARY OUTCOMES:
Breadth of the T-cell response determined as the number of reactive CD4 and CD8 T-cell epitopes to PTEg and Center for HIV/AIDS Vaccine Immunology (CHAVI) peptide set | Measured through Day 182 visit
Total magnitude of CD4 and CD8 T-cell responses measured by ICS to PTEg | Measured through Day 182 visit
Depth of the T-cell responses, determined as the variant recognition per epitope targeted by responding T cells using PTEg and CHAVI peptides | Measured through Day 182 visit
Response rate of CD4 and CD8 T-cell responses to PTEg and CHAVI peptide sets measured by ICS | Measured through Day 182 visit
Magnitude and breadth of serum neutralizing antibodies (nAbs) to a panel of standardized HIV-1 isolates | Measured through Day 364 visit
Magnitude and breadth of HIV-specific binding IgG and IgA Env antibody (Ab) responses as determined by binding Ab multiplex assay (BAMA) and peptide array | Measured through Day 182 visit

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital